CLINICAL TRIAL: NCT07244263
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Assess Efficacy and Safety of Zasocitinib in Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study of Zasocitinib in Adults With Hidradenitis Suppurativa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-HS-2001; 2025-522831-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Drug Therapy
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blinded: Zasocitinib (Dose A) (Experimental): Participants will receive zasocitinib (Dose A) from Day 1 to Week 16 during the double-blind period.
  Interventions: Drug: Zasocitinib (Dose A)
- Double-blinded: Placebo (Placebo Comparator): Participants will receive placebo from Day 1 to Week 16 during the double-blind period.
  Interventions: Other: Placebo
- Open-label: Zasocitinib (Dose A) (Experimental): Participants will receive zasocitinib (Dose A) from Week 16 to Week 52 during the open label period.
  Interventions: Drug: Zasocitinib (Dose A)

INTERVENTIONS:
Drug: Zasocitinib (Dose A) — Zasocitinib.
  Other Names: TAK-279; NDI-034858
  Arms: Double-blinded: Zasocitinib (Dose A); Open-label: Zasocitinib (Dose A)
Other: Placebo — Placebo.
  Arms: Double-blinded: Placebo

SUMMARY:
Hidradenitis Suppurativa (HS) is a skin condition that causes deep, painful bumps on the skin. These bumps usually appear in an area where the skin rubs together. They start as small bumps but may become swollen and red over time. If they fill with pus, these lumps are called abscesses; these can also burst. Over time, the area can get scars and tunnels on or under the skin. Recent studies suggest that the condition may start when hair follicles become damaged and blocked. This impacts the skin and may activate the body's germ-fighting (immune) system. This allows bacteria to grow on the skin which worsens the condition and can cause abscesses.

The main aims of this study are to learn how safe zasocitinib is, how well it works and how well adults with HS tolerate it compared with a placebo.

The participants will receive the study treatment (either zasocitinib or placebo) for up to 4 months (16 weeks). The placebo looks like the zasocitinib capsule but does not have any medicine in it. After the first 4 months, all participants (also those who initially received placebo) will then receive zasocitinib for up to 8 months (36 weeks).

During the study, participants will visit their study clinic 12 times.

ELIGIBILITY:
Inclusion Criteria:

Participant Willingness:

1. Participant is willing and able to understand and fully comply with all trial procedures and requirements (including the use of digital tools and applications), in the opinion of the investigator.
2. Participant has provided written informed consent and any required privacy authorization before the initiation of any trial procedures.

   Disease Characteristics:
3. Participants must have signs and symptoms of hidradenitis suppurativa (HS) for at least 6 months prior to screening, and a diagnosis of HS (confirmed by a dermatologist) at the screening visit with stable HS signs and symptoms for 2 months before screening, as determined by the investigator through interview or medical history.
4. Participants should have HS lesions in at least 2 distinct anatomical areas, one of which must be at least Hurley Stage II or III at both screening and Day 1.
5. Participants must have a total of greater than or equal to (>=) 5 inflammatory lesions (that is, number of abscesses plus number of inflammatory nodules) at both screening and Day 1.
6. Participants must have a history of inadequate response to a previous course of oral antibiotic for treatment of HS or exhibited recurrence, intolerance, or contraindication during that course of oral antibiotic, as assessed by the principal investigator.

   Age and Reproductive Status:
7. Participant is aged >=18 years at the time of consent. In the European Union (EU)/European Economic Area (EEA), for participants aged 65 years or older, the investigator must document a favorable benefit-risk assessment to justify the participant's inclusion in the trial.
8. Participant meets the following birth control requirement:

   1. An individual with potential for pregnancy, who is now surgically sterile; OR
   2. An individual of nonchildbearing potential with laboratory confirmation of postmenopausal status; OR
   3. If sexually active with a nonsterilized individual who produces sperm, an individual with potential for pregnancy who agrees to use a highly effective method of contraception from the signing of informed consent throughout the duration of the trial.

   The use of effective contraception will be required for participants assigned male sex at birth.

   In the EU/EEA, for participants who elect to use hormonal contraception as a form of highly effective contraception, the investigator must document a favorable benefit-risk assessment to justify the participant's inclusion in the trial at screening and every 3 months during the trial.
9. For participants in the EU/EEA, the investigator must have no reason to believe that the participant would be placed at risk by participating in the trial with regard to the European Commission decision as of 10 March 2023 on measures to minimize risk of serious side effects with JAK inhibitors (EMA/142279/2023) and the UK Medicines and Healthcare products Regulatory Agency (MHRA) guideline on Janus kinase (JAK) inhibitors: new measures to reduce risks of major cardiovascular events, malignancy, venous thromboembolism, serious infections and increased mortality as of 26 April 2023.

Exclusion Criteria:

Target Disease-Related Exclusions:

1. Participant has a draining tunnel count of greater than (>) 20 at screening or Day 1.
2. Participant has any other active skin disease or condition (for example, bacterial cellulitis, Candida intertrigo, extensive condyloma) that may, in the opinion of the investigator, interfere with the assessment of HS or participant has developed a concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the trial assessments.
3. Participant has a diagnosis of sarcoidosis, systemic lupus erythematosus, or active inflammatory bowel disease.
4. Participant has a diagnosis of inflammatory conditions other than HS, including but not limited to, psoriasis, psoriatic arthritis, and rheumatoid arthritis.

   Recent/Concurrent Infectious Disease Exclusions:
5. Tuberculosis (TB):

   1. Participants have a history of active TB infection, regardless of treatment status.
   2. Participants have signs or symptoms of active TB (including, but not limited to, chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator.
   3. Participants have evidence of latent tuberculosis infection (LTBI) as evidenced by a positive QuantiFERON (QFT) result OR 2 indeterminate QFT results, and participant does not have documentation of appropriate LTBI prophylaxis or is not able or not willing to initiate appropriate LTBI prophylaxis. Participant remains eligible if there are no signs/symptoms of active TB AND documentation of no history of active TB can be provided AND (1) participant can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines) or (2) participant has a positive QFT result or 2 indeterminate QFT results but has initiated prophylaxis (appropriate in duration and type per current local guidelines) a minimum of 2 weeks prior to Day 1. In the EU/EEA, participants with evidence of LTBI, regardless of prophylaxis treatment status, must receive approval to participate in the trial from an infectious disease or other TB specialist (for example, pulmonologist).

      Note: TB prophylaxis regimens should be administered according to local guidelines; however, because of potential interactions with zasocitinib, rifampin should not be used. For isoniazid monotherapy, a minimum of 6 months should be used. TB testing should be conducted using QFT-TB Gold submitted to the central laboratory unless alternate or additional tests are required per local guidelines.
   4. Participant has had any imaging trial during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB. X-ray is required for all participants regardless of QFT-TB Gold results unless the participant has had normal chest imaging in the 6 months prior to screening.
6. Herpes infections:

   1. Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1.
   2. Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
7. Nonherpetic viral diseases:

   1. Participant has presence of hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV RNA (nucleic acid test or polymerase chain reaction [PCR]). In the EU/EEA, if the participant has total anti-HCV antibody positivity at screening but is confirmed to have no detectable HCV RNA by PCR testing, HCV RNA PCR testing will be assessed every 3 months until end of trial (EOT).
   2. Participant has presence of positive hepatitis B virus surface antigen (HBsAg), or indeterminate HBsAg, presence of HBV DNA (regardless of serology), or positive anti-hepatitis B core antibody (HBcAb) without concurrent positive HBsAb (HBcAb+ and HBsAb-). In the EU/EEA, if the participant has total anti-HBc antibody positivity at screening but is confirmed to have no detectable HBV DNA by PCR testing, the participant will repeat HBV DNA PCR testing every 3 months until the EOT; if a participant has anti-HBsAb positivity at screening but is confirmed to have no detectable HBV DNA by PCR testing, unless the participant has documented completion of the HBV vaccination series by medical history, the participant will repeat HBV DNA PCR testing every 3 months until the EOT. Note: For other countries in which there are hepatitis B screening guidelines, these can be done per local regulations or country standard of care.
   3. Participant has positive results for HIV by serology, regardless of viral load.
8. Other infectious diseases:

   1. Participant has a history of active infection or febrile illness within 10 days prior to Day 1, as assessed by the investigator.
   2. Participant has a history of symptoms suggestive of systemic or invasive infection within 30 days prior to Day 1.
   3. Participant has a history of bacterial, viral, or fungal infection that required hospitalization or treatment with intravenous (IV) antimicrobial therapy within 8 weeks prior to Day 1, or oral antimicrobial therapy within 30 days prior to Day 1.
   4. Participant has a history of chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations (except those part of the HS clinical findings)/infections or fungal infections (except ungual onychomycosis).
   5. Participant has a history of an infected joint prosthesis unless that prosthesis has been removed or replaced at least 60 days prior to Day 1.
   6. Participant has a history of opportunistic infections (for example, Pneumocystis jirovecii pneumonia, histoplasmosis, or coccidiomycosis).
   7. Participant had a bacterial infection within 60 days prior to Day 1 for which he or she did not receive treatment.

   Noninfectious Disorders Exclusions:
9. Participant has any clinically significant medical condition, evidence of an unstable clinical condition (for example, cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, neurologic, nutritional, ophthalmologic, or immunologic), or vital signs/physical/laboratory/electrocardiogram (ECG) abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of trial results. These include but are not limited to:

   1. Participant has a history of known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency, splenectomy.
   2. Participant has a history of new or unstable autoimmune disease (including but not limited to autoimmune thyroid disease, alopecia areata, lupus, Sjogren's, myasthenia gravis, or rheumatoid arthritis).
   3. Participant had a major surgery within 60 days prior to Day 1 or has a major surgery planned during the trial.
   4. Participant has unstable, poorly controlled, or severe hypertension at screening, confirmed by 2 repeat assessments.
   5. Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association criteria.
   6. Participant has a history of lymphoproliferative disease.
   7. For participants with asthma, chronic obstructive pulmonary disease, or other pulmonary illnesses, participant has been hospitalized in the past 3 months, has ever required intubation for treatment, currently requires oral corticosteroids, or has required more than 1 course of oral corticosteroids within 6 months prior to Day 1.
   8. Participant has any of the following cardiovascular disease history:

      * A new diagnosis of atrial fibrillation or an episode of atrial fibrillation with rapid ventricular response or other dysrhythmia, nonacute cardiac hospitalization (for example, pacemaker implantation), pulmonary embolism, or deep venous thrombosis within the past 6 months prior to screening.
      * Any history of cerebrovascular event, myocardial infarction, coronary stenting, or aortocoronary bypass surgery. If, however, the investigator documents there are no suitable treatment alternatives available for the participant and it has been at least 6 months since the occurrence of any such event, the participant may enroll; in the EU/EEA, investigators must document a favorable benefit-risk assessment.
   9. Participant has significant/uncontrolled psychiatric illness, in the opinion of the investigator.
   10. Participant has any lifetime history of suicide attempts, or active suicidal ideation or suicidal behavior in the past 5 years, or any diagnosis of severe depression or other unstable psychiatric condition in the last 6 months, based on: (1) medical history; or (2) Columbia-Suicide Severity Rating Scale (C-SSRS) documentation by answering "yes" to Question 4 or 5 for suicidal ideation concerning the previous 5 years before participation on the C-SSRS at screening or Day 1; or (3) is clinically deemed to have a suicide risk by the investigator, or in the opinion of the investigator, would pose an unacceptable risk to the participant's safety or impact their ability to comply with trial procedures.
   11. Participant has a score of 15 or above at screening or Day 1 on the 8-item Patient Health Questionnaire-8 (PHQ-8).
   12. Participant has a history of active substance abuse or a history of substance abuse within 12 months prior to screening.

   Laboratory/Physical Exclusions:
10. Participant has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if they participated in the trial, in the opinion of the investigator.
11. Participant has inadequate renal, hepatic, or pancreatic function before enrollment based on the following parameters:

    1. Total bilirubin (unconjugated and/or conjugated) >1.5 × upper limit of the normal range (ULN) unless the participant has known Gilbert's syndrome that can explain the elevation of bilirubin, or
    2. Serum alanine aminotransferase (ALT) or AST >3 × ULN, or
    3. Creatinine >1.5 × ULN. Note: The participant may be retested (1 time) to meet eligibility criteria at the discretion of the investigator.
    4. Estimated creatinine clearance lesser than (<)45 milliliter per minute (mL/min) based on the Cockcroft-Gault calculation.
    5. A history of chronic pancreatitis or recent acute pancreatitis (<60 days/not fully resolved).
12. Participant has any of the following laboratory values at the screening visit:

    1. Hemoglobin <9.0 gram per deciliter (g/dL) (<90.0 gram per liter [g/L]).
    2. Absolute white blood cell count <3.0 × 10^9/L (<3000/ cubic millimeters [mm^3]).
    3. Absolute neutrophil count (ANC) of <1.0 × 10^9/L (<1000/mm^3).
    4. Absolute lymphocyte count of <0.5 × 10^9/L (<500/mm^3).
    5. Platelet count <100 × 10^9/L (<100,000/mm^3).
    6. Thyroid-stimulating hormone (TSH) (>10 milli-international units per liter [mIU/L]) or free T4 or T3 outside the normal reference range. Note: Participants would be allowed to rescreen after treatment.
    7. Triglyceride level >=750 milligram per deciliter [mg/dL] (>=8.5 millimole per liter [mmol/L]).
    8. Creatine phosphokinase (CPK) > ULN. CPK may be repeated once; if repeat value is Common Terminology Criteria for Adverse Events (National Cancer Institute) (CTCAE) Grade 1 or lower (or lesser than or equal to [<=]2.5 × ULN) and no higher than the initial value, participant remains eligible. Investigators should assess the participant for modulating factors including concomitant medications or vigorous exercise that may affect CPK levels.
    9. Participant has any other significant laboratory abnormalities that, in the opinion of the investigator, might place the participant at unacceptable risk for participation in this trial.
    10. Participant does not tolerate venipuncture or inability to be venipunctured.

    Allergies and Adverse Drug Reactions Exclusions:
13. Participant has a history of significant drug allergy (such as anaphylaxis).
14. Participant has a known or suspected allergy to zasocitinib or any of its components.

    Other Exclusions:
15. Participant has a positive pregnancy test result or plans to become pregnant during the trial period, including plans to donate ova (eggs) or sperm, or participant is pregnant or lactating/nursing.
16. Participant has a history of substance abuse within 12 months prior to Day 1.
17. Participants who have given greater than 500 mL of blood or plasma within 30 days prior to screening (during a clinical trial or at a blood bank donation) or plan to donate blood during the course of the trial.
18. Participant is compulsorily detained for treatment of either a psychiatric or physical (for example, infectious disease) illness, or is committed to an institution (for example, prison) by virtue of an order issued either by judicial or administrative authorities.
19. Participant is a trial site employee, an immediate family member (for example, spouse, parent, child, sibling), or is in a dependent relationship with trial site employee who is involved in the conduct of this trial or may consent under duress.
20. In Germany, participant is incapable of giving consent or otherwise meets criteria in Sections 136 or 137 of the Verordnung zum Schutz vor der schädlichen Wirkung ionisierender Strahlung Strahlenschutzverordnung.
21. Participants with a history of malignancy within the past 5 years prior to the screening visit are excluded, EXCEPT if the malignancy was a cutaneous squamous or basal cell carcinoma, or in situ cervical cancer that has been successfully treated and is considered cured; in the EU/EEA, investigators must document a favorable benefit-risk assessment.
22. History or current status of substance use disorder and or tobacco use disorder. For participants with excessive alcohol intake or currently smoking or using chewing tobacco or with a history of long-term smoking (>=20 pack years) or chewing tobacco use, the investigator must document a favorable benefit-risk assessment to justify the participant's inclusion in the trial.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2028-02-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve 75 Percent (%) Reduction in Hidradenitis Suppurativa Clinical Response (HiSCR75) | At Week 16
  HiSCR75 is defined as at least a 75% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess or draining tunnel count relative to baseline.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve 50% Reduction in HiSCR50 | At Week 16
  HiSCR50 is defined as at least a 50% reduction in the total AN count with no increase in abscess or draining tunnel count relative to baseline.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From start of study drug up to Week 56
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a trial intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the trial intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (49):
- United States (15):
  - Mayo Clinic, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - First OC Dermatology Research, Fountain Valley, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - StracSkin, PLLC, Greenland, New Hampshire
  - Northwell Health Physician Partners, Lake Success, New York
  - Mount Sinai Doctors, New York, New York
  - Apex Clinical Research Center, LLC., Mayfield Heights, Ohio
  - ODRC Enterprises, LLC dba Oregon Dermatology and Research Center, Portland, Oregon
  - Arlington Research Center, Inc., Arlington, Texas
  - Texas Dermatology Research Center, Dallas, Texas
- Australia (5):
  - Skin & Cancer Foundation - The Skin Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Canada (8):
  - Beacon Dermatology, Calgary, Alberta
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Ryan Clinical Research Inc., Newmarket, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - DIEX RECHERCHE Quebec, Québec, Quebec
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Southern Medical Universtiy - Dermatology Hospital (SMUDH) (Guangdong Provincial Dermatology Hospital), Guangzhou, Guangdong
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology (HUST), Wuhan, Hubei
  - Huashan Hospital, Fudan University, Shanghai, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
- France (6):
  - CHU NICE, Nice, Alpes Maritimes
  - APHM, Marseille, Bouches Du Rhone
  - Cabinet medical du Docteur RUER, Martigues, PACA
  - Hopital Edouard Herriot, Lyon, Rhone
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - CHU de Rouen, Rouen
- Germany (4):
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Katholisches Klinikum Bochum gGmB, Bochum, Northrhine Westfalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz - Hautklinik und Poliklinik - Clinical Research Center (CRC), Mainz, Rhineland-Palatine
  - Charite Dermatology, Berlin
- ErasmusMC, Rotterdam, South Holland, Netherlands
- Poland (5):
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak SpAAka Partnerska, Wroclaw, DolnoAlAskie
  - Klinika Ambroziak Dermatologia, Warsaw, Masovia
  - PaAstwowy Instytut Medyczny MSWiA, Warsaw, Mazowsze
  - Klinika Dermatologii, Uniwersytecki Szpital Kliniczny, Rzeszów, Podkarpackie, Poland
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp z o.o., Malbork, Pomeranian

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/57d8039b3c094c40??page=1&idFilter=TAK-279-HS-2001